CLINICAL TRIAL: NCT06589193
Title: Comparison of the Clinical and Microbiological Effects of CHX and HOCl Containing Mouthwashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Mehtap Bilgin Çetin, Director, Baskent University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MR1234
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dental Plaque
Keywords: Hypochlorous acid; chlorhexidine gluconate; antiplaque; anti-inflammatory; gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: 4-day plaque regrowth study model
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HOCl (Experimental)
  Interventions: Other: HOCl
- CHX (Active Comparator)
  Interventions: Other: CHX

INTERVENTIONS:
Other: HOCl — 10ml,twice a day
  Arms: HOCl
Other: CHX — 10ml,twice a day
  Arms: CHX

SUMMARY:
The primary objective of the study is to compare the antiplaque and anti-inflammatory effects of HOCl mouth rinse with those of CHX mouth rinse. The secondary objective is to evaluate and compare the antimicrobial activities of HOCl mouth rinse and CHX mouth rinse on dental biofilm.

DETAILED DESCRIPTION:
The primary objective of the current clinical study is to compare the antiplaque and anti-inflammatory efficacy of HOCl mouth rinse with that of CHX mouth rinse. The secondary objective is to compare the antimicrobial activities of these two mouth rinses on dental biofilm. This single-center, triple-blind, randomized controlled crossover study was completed with 26 participants. In the study, the same participants used both HOCl (0.02%) and CHX (0.2%) mouth rinses over a 4-day re-plaque formation model. Following each mouth rinse usage, supragingival dental plaque biofilm samples were collected, and clinical parameters including the Modified Plaque Index, Bleeding on Probing Index, and Modified Stain Index were recorded. Additionally, participants were asked to evaluate the mouth rinses they used via a questionnaire. In conclusion, HOCl mouth rinse has demonstrated antiplaque efficacy comparable to that of CHX mouth rinse. When evaluating total bacterial counts, both mouth rinses exhibited similar antimicrobial effectiveness. Within the limitations of this study, HOCl may be considered a promising antimicrobial agent for dental plaque control.

ELIGIBILITY:
Inclusion Criteria:

* Being systematically healthy
* Having at least 22 natural teeth (236)
* Not smoking
* Participants must not drink alcohol and must work during their term

Exclusion Criteria:

* Having periodontitis and gingivitis
* Being breastfeeding or pregnant
* Using medication that may affect periodontal status
* Having used antibiotics in the last month
* Having used any mouthwash in the last month
* Using fixed, removable dentures or orthodontic appliances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
plaque index | 1 month
  Plaque index results were evaluated regionally and full mouth for CHX and HOCl groups.

SECONDARY OUTCOMES:
microbiology | 1 month
  Microbiological data were evaluated on plaque samples taken from molar teeth for CHX and HOCl groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Bilgin Cetin, Assoc. prof., Principal Investigator — Başkent Üniversitesi
Locations (1):
- Baskent University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lafaurie GI, Zaror C, Diaz-Baez D, Castillo DM, De Avila J, Trujillo TG, Calderon-Mendoza J. Evaluation of substantivity of hypochlorous acid as an antiplaque agent: A randomized controlled trial. Int J Dent Hyg. 2018 Nov;16(4):527-534. doi: 10.1111/idh.12342. Epub 2018 Apr 2. PMID 29608039